CLINICAL TRIAL: NCT02786394
Title: REACH Lifestyle Program for Older Adults
Brief Title: Return to Everyday Activities in the Community and Home
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Maureen C. Ashe, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H16-00670
Record Dates: First submitted 2016-05-18; First posted 2016-06-01 (Estimated); Results first posted 2022-04-20 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Aging; Activity; Lifestyle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- REACH Participant Course (Experimental): This study will run twice a week over 6 weeks with 6 REACH sessions optional walking program sessions. The optional walking program will be run by SportMedBC and may consist of one or more educational sessions (e.g., nutrition). Each REACH session introduces new topics, strength and balance activities and home practices which progressively build on each other. We will ask participants to provide feedback after each session, and in two to three 30 minutes recorded interviews (in-person or over the telephone) at the end of the study.
  Interventions: Behavioral: REACH

INTERVENTIONS:
Behavioral: REACH — REACH is a lifestyle intervention program which aims to reduce sedentary behaviour, increase physical activity, and increase strength and balance. The REACH program is comprised of six sessions which include evidence-based education, behaviour change theory, and activity instruction. REACH also teaches goal setting techniques, mindfulness, and encourages active community engagement. In this study we are running the REACH program for women aged 55 and older alongside a supplementary optional walking program run by SportMedBC.

SUMMARY:
The purpose of this study is to test feasibility for the delivery and perceptions of a lifestyle model for middle-aged and older adults by involving participants in its development. The goal of the program is to reduce sedentary behaviour, increase physical activity, and increase strength and balance. An optional walking program will be run in parallel to emphasize the importance of moving more. Participants will be asked to fill out questionnaires on course delivery, content and effect throughout the program and 2-3 recorded interviews throughout the study. We will collect measurements of physical performance before and after the program.

DETAILED DESCRIPTION:
This study aims to describe the delivery of a lifestyle model for older adults. Return to Everyday Activities in the Community and Home (REACH) is a health promotion program aimed at middle-aged and older adults. The goal of REACH is to reduce sedentary behaviour, increase physical activity, and increase strength and balance. The REACH program is comprised of six sessions which include evidence-based education, behaviour change theory, and activity instruction. REACH also teaches goal setting techniques, mindfulness, and encourages active community engagement. In this study we are running the REACH program for women aged 55 and older alongside a supplementary optional walking program run by SportMedBC. We will gather pre- and post-intervention measures of program perceptions, delivery psychological variables and physical performance outcomes. We will also collect participant feedback about course delivery, content and effect throughout the program. This study will allow us to describe the delivery strategies of REACH and involve the participants in the development of the REACH program. The optional walking program will emphasize the importance of increasing daily physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Participants included will be women aged 55 and older.
* Participants must speak English.
* Participants must be able to walk a minimum of four city blocks, climb a flight of stairs and take part in a physical activity and walking program.
* Participants must be cleared by a health care professional to participate using the Physical Activity Readiness Questionnaire for Everyone (Par-Q+) assessment to determine if they are physically able to take part in the activity program.

Exclusion Criteria:

* Individuals will be excluded if they are men, under the age of 55 and/or do not speak English.

Ages: 55 Years to 105 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Ashe, PhD, Principal Investigator — University of British Colubia
Locations (1):
- Centre for Hip Health and Mobility, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashe MC, Edwards NY, Taylor A, Burnett L, Giangregorio L, Milne K, Clemson L, Fleig L. Return to Everyday Activity in the Community and Home: a feasibility study for a lifestyle intervention to sit less, move more, and be strong. Pilot Feasibility Stud. 2019 Jun 28;5:84. doi: 10.1186/s40814-019-0467-9. eCollection 2019. PMID 31297236

RESULTS

PARTICIPANT FLOW:
Groups:
- REACH Participant Course: This study will run twice a week over 6 weeks with 6 REACH sessions and optional walking program sessions. The optional walking program will be run by SportMedBC and may consist of one or more educational sessions (e.g., nutrition). Each REACH session introduces new topics, strength and balance activities and home practices which progressively build on each other. We will ask participants to provide feedback after each session, and in two to three 30 minutes recorded interviews (in-person or over the telephone) at the end of the study.
  REACH: REACH is a lifestyle intervention program which aims to reduce sedentary behaviour, increase physical activity, and increase strength and balance. The REACH program is comprised of six sessions which include evidence-based education, behaviour change theory, and activity instruction. REACH also teaches goal setting techniques, mindfulness, and encourages active community engagement. In this study we are running the REACH program for women aged 55 and older alongside a supplementary optional walking program run by SportMedBC.
Period: Overall Study
Arm/Group | REACH Participant Course
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [57.5 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 11

OUTCOME MEASURES:

1. Primary Outcome: REACH Session Feedback
Description: We will ask participants to report feedback and experience following each REACH session. As this was a pilot study we wanted to capture participants' perceptions of the program. When appropriate, we adjusted the content/delivery in consultation with participants. We also asked participants to rate their overall experience with REACH [1 (low) - 7 (high)].
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 10
score on a scale | 5.94 (0.59)

2. Secondary Outcome: Physical Activity Identity
Description: A questionnaire will be administered at the beginning and end of the REACH sessions to determine how the participant identifies themselves with regard to physical activity. The minimum score is 9 and the maximal score is 63; the higher the score the better.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 10
score on a scale | 46.2 (10.5)

3. Secondary Outcome: Grit Score
Description: A questionnaire will be used to determine how the participant perceives their ability to stick with (follow through on) projects or goals. The higher the score the better. Scores range from 1 (not like me to) to 5 (very much like me).
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 10
score on a scale | 4.1 [3.4 to 4.5]

4. Secondary Outcome: Automaticity Subscale of the Self-Report Habit Index
Description: A questionnaire will be administered to determine the participant's level of automaticity for physical activity. Scores are based on a 7-point Likert scale (1=strongly disagree- 7=strongly agree). In other words, participants rate how "automatic" their behavior is for physical activity.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 10
score on a scale | 4.9 (1.6)

5. Secondary Outcome: Sedentary Behaviour
Description: We will request participants record their sedentary behaviour data from activity monitors.
Time Frame: weekly for 6 weeks
Population: Not able to use data due to reporting issues.
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 0

6. Secondary Outcome: Hourly Activity
Description: We will request participants to record their hourly activity (number of hours active per day) data from activity monitors.
Time Frame: weekly for 6 weeks
Population: unable to collect data
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 0

7. Secondary Outcome: Step Count
Description: We will request participants to record their daily step count data from activity monitors.
Time Frame: weekly for 6 weeks
Measure: Median (Inter-Quartile Range); unit: steps/day
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 8
steps/day | 7954 [6861 to 11,401]

8. Secondary Outcome: Number of REACH Sessions Attended
Description: Number of REACH sessions attended during the project.
Time Frame: weekly for 6 weeks
Measure: Mean (Standard Deviation); unit: Sessions attended
Units Other Than Participants: Sessions
Arm/Group | REACH Participant Course
Number analyzed (Participants) | 10
Number analyzed (Sessions) | 6
Sessions attended | 5 (1)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- REACH Participant Course: This study will run twice a week over 8 weeks with 6 REACH sessions 8 optional walking program sessions. The optional walking program will be run by SportMedBC and may consist of one or more educational sessions (e.g., nutrition). Each REACH session introduces new topics, strength and balance activities and home practices which progressively build on each other. We will ask participants to provide feedback after each session, and in two to three 30 minutes recorded interviews (in-person or over the telephone) at the end of the study.
  REACH: REACH is a lifestyle intervention program which aims to reduce sedentary behaviour, increase physical activity, and increase strength and balance. The REACH program is comprised of six sessions which include evidence-based education, behaviour change theory, and activity instruction. REACH also teaches goal setting techniques, mindfulness, and encourages active community engagement. In this study we are running the REACH program for women aged 55 and older alongside a supplementary optional walking program run by SportMedBC.
Arm/Group | REACH Participant Course
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No